CLINICAL TRIAL: NCT07123753
Title: EFFECTS OF CLASSICAL FOOT EXERCISES AND FOOT CORE EXERCISES ON PAIN, BALANCE, GAIT AND LOWER EXTREMITY PERFORMANCE IN ADOLESCENTS WITH PES PLANUS
Brief Title: Exercises for Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Aysel TOPÇU, Physiotherapist, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GISTU-FTR-AT-1; GISTU-FTR (Other: GISTU)
Record Dates: First submitted 2025-03-12; First posted 2025-08-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pes Planus
Keywords: Adolescent, foot core exercise, foot classic exercise, pes planus
MeSH Terms: conditions — Flatfoot | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator): CLASSIC FOOT EXERCISE WILL BE APPLIED
  Interventions: Other: EXERCİSE
- WORKING GROUP (Active Comparator): CORE FOOT EXERCISE WILL BE APPLIED
  Interventions: Other: EXERCİSE

INTERVENTIONS:
Other: EXERCİSE — The aim of this study is to examine the effects of classical foot exercises and foot core exercises on pain, balance, gait and lower extremity performance in adolescents with pes planus. This study is planned to be a randomized controlled trial. Participants will be randomly divided into 2 groups. Classic foot exercises will be applied to individuals in the classical foot exercises group for 12-15 minutes, and foot core exercises will be applied to individuals in the core exercises group for 12-15 minutes twice a week for a total of 8 weeks. Pes planus status of individuals included in the study will be evaluated with the navicular drop test. Pain will be evaluated with the foot function test, balance with the star balance test, gait analysis with the footprint method and lower extremity muscle performance with the functional muscle strength assessment for individuals in both groups before and after the application. The evaluations will be applied face to face by the same physiotherapi

SUMMARY:
Pes planus is a musculoskeletal syndrome in which the medial longitudinal arch (MLA) of the foot is reduced or flattened. It results from a combination of static and dynamic abnormalities. Various predisposing factors such as increased weight, foot injury, and musculoskeletal disorders are associated with this problem. In addition, studies have emphasized that there is a significant relationship between abnormal foot posture and gait mechanics.

DETAILED DESCRIPTION:
Pes planus is a musculoskeletal syndrome in which the medial longitudinal arch (MLA) of the foot is reduced or flattened. It results from a combination of static and dynamic abnormalities. Various predisposing factors such as increased weight, foot injury, and musculoskeletal disorders are associated with this problem. It has been reported that pes planus is associated with various disorders seen in the lower extremity such as patellofemoral pain syndrome and medial tibial stress syndrome. In addition, studies have emphasized that there is a significant relationship between abnormal foot posture and gait mechanics. Therefore, our aim in this study is to examine the effects of classical foot exercises and foot core exercises on pain, balance, gait, and lower extremity performance in adolescents with pes planus. This study is planned to be a randomized controlled trial. Participants will be randomly divided into 2 groups. Individuals in the classical foot exercises group will be subjected to classical foot exercises for 12-15 minutes, and individuals in the core exercises group will be subjected to foot core exercises for 12-15 minutes twice a week for a total of 8 weeks. Individuals included in the study will be assessed for pes planus status with the navicular drop test. For both groups, pain will be assessed with the foot function test, balance with the star balance test, gait analysis with the footprint method, and lower extremity muscle performance with functional muscle strength assessment, before and after the application. The assessments will be applied face to face by the same physiotherapist to all group members.

ELIGIBILITY:
Inclusion Criteria:

Those who have not had any surgery in the last 6 months

Individuals who do not have any physical or mental disabilities

Individuals who volunteer to participate in the study

Exclusion Criteria:

Individuals with major foot deformities other than pes planus Individuals with any physical or mental disability Individuals with a history of lower extremity injury in the last 6 months

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
The navicular drop test | Change from Baseline at 8 weeks
  The navicular drop test is a test used in the clinic to determine the presence and degree of pes planus. It will be used to distinguish participants with and without pes planus.). In this test, first the navicular tubercle is palpated and marked, and the distance between the navicular tubercle and the floor is measured with a ruler while the person is in a sitting position and the feet are only in contact with the floor (without putting weight on the feet). Then the person stands up and puts equal weight on their feet, and the distance between the navicular tubercle and the floor is measured again. Measurements are made bilaterally and recorded in millimeters (mm) or centimeters (cm). In the navicular drop test, the difference between the weighted and unweighted measurements is considered normal (neutral) between 5-9 mm, excessive pronation of 10 mm and above, and excessive supination of 4 mm and below.
STAR BALANCE TEST | Change from Baseline at 8 weeks
  Star balance test (SBT) is one of the tests frequently used to evaluate lower extremity dynamic balance and postural control. SBT is a test that measures the maximum extension an individual can achieve by maintaining balance and performing a single-leg squat on lines drawn at 45-degree intervals in eight different directions.
The foot function index | Change from Baseline at 8 weeks
  The foot function index is a test used to determine pain, disability and activity limitation. It is a scale consisting of a total of three parameters and 23 items. The pain subscale contains nine items and measures the severity of foot pain in different situations. The disability subscale contains 9 items and evaluates the severity of the difficulty in performing functional activities due to the person's foot problems. The activity limitation subscale contains 5 items and measures the person's activity limitations due to foot problems. The AFI is a scale filled out by the person himself. A high score indicates more pain, disability and activity limitation.
Gait Assessment (Footprint method): | Change from Baseline at 8 weeks
  Gait Assessment (Footprint method): General gait parameters are temporal and distance factors, cycle time (cadence), step length and speed. These are the simplest form of objective gait assessment. Only a stopwatch, a tape measure and some talcum powder are required. The individual will be asked to walk naturally and will be allowed to stand on their own feet. The individual will step on a tray of talcum powder and then will be asked to walk across a black bag. The left and right step lengths, step length, toe angle and an idea of the foot contact pattern are obtained.
Dynamic Gait Index | Change from Baseline at 8 weeks
  The Dynamic Gait Index (DGI) is a clinical measure that assesses the ability of a person to adapt to complex walking tasks commonly encountered in daily life. The DGI is based on a person-environment mobility disability model in which environmental demands are categorized as distance, time, environment, terrain, physical load, attention, postural transitions, and intensity, and represents the external demand that must be met for an individual to move in a given environment. Item 1 of the DGI is considered the reference or baseline task and examines the ability to walk under low-intensity conditions (self-paced, level-surface walking). The remaining 7 items examine the person's ability to adapt their gait to task demands in 4 environmental dimensions.Each item is scored on an ordinal scale (0-3) based on gait pattern, speed, and assistance level, with total scores ranging from 0 (worst) to 24 (best)."
Functional Muscle Strength Evaluation | Change from Baseline at 8 weeks
  Functional Muscle Strength Evaluation: The number of repetitions of the movement in a certain period of time is a valid and reliable method used effectively in functional muscle strength evaluation. In our study, individuals' lower extremity functional muscle strength will be evaluated with a 30-second maximum repetition test. Within the scope of this evaluation, individuals are asked to perform 3 closed kinetic chain exercises involving large muscle groups for standing and walking. These are (1) "Lateral Step-up" test (taking a side step to a 20 cm bench), (2) "Sitto-Stand" test (standing up without sitting without using the arms), (3) "Attain Stand Through Half Knee" (moving from kneeling position to half kneeling position) test. The maximum number of repetitions the person does in 30 seconds is noted. A higher number of repetitions indicates better functional performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Nizip, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No